CLINICAL TRIAL: NCT06907095
Title: A Prospective Cohort to Evaluate the Ability of Different Body fLuid-derived Approaches to Detect EArly-stage Cancers Among High-risk Individuals
Brief Title: Cohort Evaluation of Body Fluids Early Detection of Cancer in High-risk Individuals
Acronym: LEAH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-A02283-44; 2023/3648 (Other: CSET number (Gustave Roussy ID))
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Risk of Breast Cancer; Risk of Gynaecological Cancer; Risk of Colorectal Cancer; Risk of Upper Gastrointestinal Cancers; Risk of Hepatic Cancers; Risk of Lung Cancer; Risk of Skin Cancers Except Basal-cell Carcinomas; Risk of Head and Neck Cancers; Risk of Mesothelioma; Risk of Kidney Cancer; Risk of Prostate Cancer; Risk of Urothelial Cancers; Risk of Endocrine Cancers; Risk of Hematologic Malignancies; Risk of Several Cancer Types; Risk of Second Malignancy in Individuals Treated for a Childhood Cancer; Risk of Neoplasia
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: 2 cohorts: individuals at high risk of invasive cancer and individuals at low risk of invasive cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individuals at low risk of invasive cancer (Active Comparator): A cohort of individuals who are not considered at increased risk (low risk) of cancer seen in consultation for a problem defined as benign will also be recruited and be used for certain secondary and exploratory objectives.
  Interventions: Diagnostic Test: biological samples
- individuals at high risk of invasive cancer (Active Comparator): Individuals with an estimated risk ≥ 4% of occurrence of any invasive cancer or malignancy (except for basal cell carcinoma of the skin) in the following three years after inclusion will be proposed the trial. This 4% cumulative risk represents the addition of i. the participant's general risk of any cancer or malignancy based on her/his age and ii. her/his risk of a specific malignancy based on her/his risk profile.
  Interventions: Diagnostic Test: biological samples

INTERVENTIONS:
Diagnostic Test: biological samples — biological samples (blood, urine, saliva)

SUMMARY:
LEAH is a prospective, observational, single-centre, non-randomised, open-label study of people at increased risk of cancer or malignant disease.

The main objective of LEAH is to evaluate and compare the sensitivity of different tests on body fluids to detect cancers that will occur within 3 years of inclusion in the study, in a cohort of individuals identified as being at increased risk of cancer.

ELIGIBILITY:
Inclusion Criteria increased risk cohort:

1. Are aged 18 or more
2. Have a cumulative 3-year risk of developing any cancer ≥ 4% (including the situation specific cancers + other cancers) defined as follows:

   1. Situations at increased risk of breast cancer

      * Women carrying germline pathogenic (P) or likely pathogenic (LP) variants of BRCA1, BRCA2, TP53, PALB2, PTEN, CDH1 genes without prophylactic mastectomy, aged ≥ 40 years, or
      * Men with germline (P) or (LP) variants in the BRCA2 gene, aged ≥ 40 years, or
      * Women with a personal history of an histological atypical breast lesion in the past 5 years and aged ≥ 50 years, or
      * Women with a personal history of unilateral breast cancer (including ductal carcinoma in situ) diagnosed more than 5 years before inclusion, and currently aged ≥ 60 years, or
      * Women who received chest radiotherapy before age 30 years and currently aged ≥ 25 years, or
      * Women with an invasive breast cancer risk > 2.5% over the next 5 years, as defined by risk scores +/- genotyping, and aged ≥ 50 years, or
      * Individuals identified at increased risk in MyPeBS trial (> 2.5% over the next five years) (www.mypebs.eu) can be eligible for the study, if aged ≥ 50 years, or
   2. Situations at increased risk of gynaecological cancer

      * Women with a Lynch syndrome - germline (P) or (LP) variants in hMLH1, MSH2, hMLH6, PMS2, and aged ≥ 30 years, or
      * Women carrying germline (P) or (LP) variants of BRCA1, BRCA2, PALB2, RAD51C or RAD51D, PTEN genes without prophylactic oophorectomy, aged ≥ 40 years, or POLE and POLD1, and aged > 30 years; or SMARCA4 or DICER1 and aged > 18 years or
   3. Situations at increased risk of colorectal cancer

      * Men or women with a Lynch syndrome - germline (P) or (LP) variants in hMLH1, MSH2, hMLH6, PMS2, APC, POLE, POLD1, BMPR1A, SMAD4 or biallelic MuTYH genes, and aged ≥ 40 years, or
      * Individuals with an increased risk of colorectal cancer defined by the following criteria and aged ≥ 50 years, or
      * First-degree relative diagnosed with colorectal cancer before the age of 60 years, or
      * Two or more 1st degree relatives diagnosed with colorectal cancers at any age, or
      * Personal history of any colorectal adenoma before the age of 50 years or adenomatous polyps > 1 cm, villous adenomas, dysplastic adenomas, or ≥ 3 adenomatous polyps after the age of 50 years, or
      * Inflammatory Bowel Disease (Crohn's Disease; Ulcerative Colitis) after the age of 50 years, or
   4. Situations at increased risk of upper gastrointestinal cancers

      * Carriers of an STK11 or CDH1 germline (P) or (LP) variants and aged > 30, or
      * Individuals with an increased risk of esophageal adenocarcinoma: Barrett's esophagus with high-grade dysplasia, or
   5. Situations at increased risk of hepatic cancers

      - Individuals at increased risk of hepatocellular carcinoma because of documented liver fibrosis or cirrhosis (whether secondary to non-alcoholic steatohepatitis, alcohol-related, or virus-related), or
   6. Situations at increased risk for pancreatic cancers

      * Patients with a family history with > 2 pancreatic cancers in close relatives and aged >50 or
      * Chronic pancreatitis and aged >50 or carriers of PRSS1 or SPINK1 germline (P) or (LP) variants or
      * Patients at increased risk of pancreatic cancer based on a composite score or
      * Carriers of CDKN2A germline (P) or (LP) variants or
      * Carriers of germine (P) or (LP) variants in BRCA2, ATM, BRCA1, PALB2, or Lynch syndrome-associated gene alterations with a first-degree or multiple family history of pancreatic ductal carcinoma (PDAC) or
      * Patients with a Peutz-Jeghers syndrome (STK11 germline (P) or (LP) variants) or
   7. Situations at increased risk of lung cancer

      - History of heavy smoking > 20 pack-years among active or previous smokers who have quitted up to 10 years ago, and aged ≥ 50 years, or
   8. Situations at increased risk of skin cancers except basal-cell carcinomas

      * Carriers of germline (P) or (LP) variants in CDKN2A/CDK4 or BAP1 genes, aged ≥ 50 years or
      * Carriers of germline (P) or (LP) variants of genes that predispose to skin cancers (Xeroderma pigmentosum, etc…) or
   9. Situations at increased risk of head and neck cancers

      * Individuals with high-grade dysplasia or carcinoma in situ of the upper aero digestive tract within the last 10 years, and aged ≥ 50 years, or
      * Individuals with oral lichen planus diagnosed more than 10 years ago, and aged ≥ 50 years or
      * Previous history of a head and neck cancer in complete remission for ≥ 5 years, aged ≥ 50 years, and at least one of the following criteria:

      Current or former smoker > 10 pack-years Current or former alcohol consumption > 14 units/week
   10. Situations at increased risk of mesothelioma

       - Individuals with a history of relevant professional exposure to asbestos, and/or germline (P) or (LP) variants in BAP1, and aged ≥ 50 years, or
   11. Situations at increased risk of kidney cancer

       - Carriers of germline (P) or (LP) variants in the BAP1, VHL, FH, cMET, FLCN, SDH-B genes, and aged ≥ 50 years, or
   12. Situations at increased risk of prostate cancer

       * Men aged ≥ 40 year with any of the following:
       * Strong family history: a first- or second-degree relative with metastatic prostate cancer, ovarian cancer, male breast cancer, female breast cancer aged ≤ 45 years, colorectal or endometrial cancer aged ≤ 50 years, pancreatic cancer or two or more first- or second-degree relatives with breast, prostate (but not clinically localized grade group 1), colorectal or endometrial cancer at any age, or
       * Carriers of germline (P) or (LP) variants in BRCA1, BRCA2, ATM, HOXB13, hMLH1, MSH2, hMLH6, and PMS2, and aged > 45
   13. Situations at increased risk of urothelial cancers

       * History of heavy smoking > 30 pack-years, among active or previous smokers who have quitted up to 10 years ago, and aged ≥ 50 years, or
       * Lynch syndrome with a germline (P) or (LP) variants in hMLH1, MSH2, hMLH6, PMS2, and aged ≥ 40 years, or
   14. Situations at increased risk of endocrine cancers

       * Increased risk of pheochromocytoma paraganglioma in individuals with germline (P) or (LP) variants in RET, VHL, SDHB, SDHD, and aged ≥ 35 years, or
       * Multiple endocrine neoplasia syndrome in individuals with germline (P) or (LP) variants in RET or MEN1, and aged ≥ 40 years, or
   15. Situations at increased risk of hematologic malignancies

       * Individuals aged ≥ 50 years with any of the following:
       * Clonal hematopoiesis of indeterminate potential, or
       * Aplastic anemia, or
       * Predisposing genetic alterations (P) or (LP) variants in GATA2, RUNX1, ANKRD26, ETV6, TP53, CEBPA, or DDX41 genes, or copy number variation of chromosome 14q32 region (CNVdup14), or
       * Patients who received high doses of platinum or other compounds who are estimated to have a > 2% risk of secondary hematological malignancies at 3 years, or
   16. Situations at increased risk of several cancer types

       * Germline deleterious mutations of TP53 (Li-Fraumeni syndrome), and aged > 18 or
       * Germline deleterious (P) or (LP) variants in PTEN, Cowden syndrome, and other PTEN-opathies, aged ≥ 30 years, or
       * Personal history of allogenic organ transplantation at least five years before the inclusion, with long-term ongoing immunosuppressive treatment, and aged ≥ 50 years, or
       * Chronic HIV carriers aged > 50, or
   17. Situations at increased risk of second malignancy in individuals treated for a childhood cancer

       * Brain radiation therapy during childhood, and aged ≥ 18 years, or
       * Childhood malignancy which required chemotherapy and/or radiation therapy, and aged ≥ 40 years, or
3. Beyond the situations described previously, the following individuals are also eligible for LEAH:

   1. Increased risk of neoplasia linked to an underlying professional exposure, with a specific cancer risk estimated to be at least 2 % at 3 years, and aged ≥ 50 years, or
   2. Other situation: Any particular situation with accumulation of several risk factors likely to induce cancer with a specific risk of cancer estimated at least 2% at 3 years.
4. Participants with a personal cancer or hematological malignancy history are allowed if they are in complete remission at least 5 years from the primary diagnosis
5. All participants must understand spoken and written French language,
6. All participants must agree to comply with the protocol requirements,
7. All participants must understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
8. All participants must be able to access internet through their telephone or a computer

Inclusion criteria, control group

1. Individuals seen for a rapid diagnostic procedure at the center as part of the Instadiag programme, that led to a diagnosis of a benign condition
2. Who do not have a high risk situation as defined previously
3. Agree to participate
4. Aged >18
5. They must understand spoken and written French language,
6. They must agree to comply with the protocol requirements,
7. They must understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
8. They must be able to access internet through their telephone or a computer

Exclusion Criteria:

1. Known prior diagnosis of cancer or hematological malignancy within the past 5 years except for non-melanoma skin cancers, in situ cervical cancers and for patients with germline TP53 alterations,
2. Presence of signs or symptoms of cancer at enrolment,
3. Acute exacerbation of an autoimmune condition requiring escalation in medical therapy within 14 days prior to enrolment,
4. Any medical condition with a high likelihood of mortality within three years,
5. Physical or psychological conditions considered not to be compatible with the study and not likely to comply with follow up requirements,
6. Individuals under guardianship or deprived of their liberty by a judicial or administrative decision or incapable of giving their consent,
7. Women carriers of (P) or (LP) variants in BRCA1, BRCA2, PALB2, gene considering prophylactic mastectomy in a near future or aged less than 40 years (since their absolute risk of cancer is lower than the expected threshold)
8. Received a blood transfusion within the last week before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5909 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
sensitivity of techniques derived from body fluids in the detection of any invasive cancer | baseline and In case of cancer within 3 years
  The primary endpoint is the sensitivity of body fluid-derived techniques in the detection of any invasive cancer (except for non-melanoma skin cancers) in the 36 months period following body fluid collection among individuals at increased risk of cancer.

SECONDARY OUTCOMES:
Evaluation of the 3-year early detection performance of techniques derived from body fluids | baseline and In case of cancer within 3 years
  for different evaluation criteria: < stage 2 cancer, any invasive cancer (SO.1, SO.2 and SO.3). These performances will be evaluated in individuals at increased risk of cancer and in subgroups of individuals with several cancer-specific risk situations, using standard performance indices (sensitivity, specificity, precision, negative/positive predictive value, accuracy, etc.) corrected for censoring.
Evaluation in terms of predicting the risk of developing invasive cancer of the added value at 3 years of body fluid-derived techniques and their various combinations compared with standard baseline factors | baseline and In case of cancer within 3 years
Assessment of the ability of body fluid-derived techniques to identify the tissue of origin by agreement between the location predicted by the body fluid-derived techniques and the tissue of origin. | baseline and In case of cancer within 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Delaloge, MD, Study Chair — Gustave Roussy, Veillejuif, France
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No